CLINICAL TRIAL: NCT03646682
Title: Pharmakokinetik of Caffeine in Epiretinal Membranes After Oral Intake: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department of Ophthalmology, Professor, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CaffERM
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Vitrectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine group (Experimental): 180mg of caffeine will be given orally one jour before vitrectomy with membrane peeling
  Interventions: Procedure: vitrectomy with membrane peeling
- control group (Active Comparator): no caffeine will be given before vitrectomy with membrane peeling, patients are drinking no coffee in general
  Interventions: Procedure: vitrectomy with membrane peeling

INTERVENTIONS:
Procedure: vitrectomy with membrane peeling — during vitrectomy with membrane peeling a prob of the vitreous body and the excised epiretinal membrane will be harvested for gas-chromatography/mass spectrometry

SUMMARY:
Caffeine concentrations in the vitreous Body and exzised epiretinal membranes are measured by gas-chromatography/mass spectrometry.

DETAILED DESCRIPTION:
Caffeine concentrations in the vitreous Body and exzised epiretinal membranes are measured by gas-chromatography/mass spectrometry. One hour before surgery patients in the caffeine Group will receive 180mg of caffeine. in all patients vitrectomy with Membrane Peeling will be performed, due to epiretinal membranes

ELIGIBILITY:
Inclusion Criteria:

* epiretinale membrane

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
concentration of caffeine in vitreous probes and epiretinal membranes | one hour
  concentration of caffeine in the probes will be measuread by gas-chromatography/mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Professor, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria